CLINICAL TRIAL: NCT05972889
Title: Randomized Blinded Evaluation of the Effects of Transcutaneous Electrical Nerve Stimulation and Interferential Current Compared to a Sham Device and Standard of Care in Patients With Non-Specific Chronic Lower Back Pain
Brief Title: Randomized Blinded Evaluation of the Effects of TENS and IFC Compared to a Sham Device and SOC in Patients With Non-Specific CLBP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zynex Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ZMI-2023-NexWave-vs-Sham
Record Dates: First submitted 2023-07-25; First posted 2023-08-02 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Non-Specific Chronic Lower Back Pain
Keywords: TENS; IFC

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (5):
- Device TENS (Experimental)
  Interventions: Device: NexWave
- Device IFC (Experimental)
  Interventions: Device: NexWave
- Sham TENS (Sham Comparator)
  Interventions: Device: Sham
- Sham IFC (Sham Comparator)
  Interventions: Device: Sham
- Control (No Intervention): Subjects continue with current standard of care only for 4 weeks with the option to crossover to the NexWave Device group for an additional 4 weeks (up to 8 total weeks).

INTERVENTIONS:
Device: NexWave — Device subjects receive designated treatment mode twice daily for up to 8 weeks.
  Arms: Device IFC; Device TENS
Device: Sham — Sham subjects provided with Sham Device and treatment instructions identical to that of NexWave Device Arm for their designated Sham Arm. Sham subjects participate for 4 weeks with the option to crossover to the NexWave Device Arm for an additional 4 weeks (up to 8 weeks total).
  Arms: Sham IFC; Sham TENS

SUMMARY:
This is a prospective, sham-controlled, randomized, single-blinded, multi-center study comparing two different modes of the NexWave device, transcutaneous electrical nerve stimulation (TENS) and interferential current (IFC), with an identical non-functioning NexWave sham device or self-defined standard of care for improvement of pain intensity of non-specific CLBP.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-70, or older if specified by law
* Non-specific chronic lower back pain defined as:

  1. Having lasted ≥3 months in duration
  2. Current Visual Analogue Scale (VAS) pain rating ≥50 out of 100 (or an equivalent of 5 out of 10 on a 10-point scale)
  3. No radiating pain below the knee
  4. ≥75% back or buttock pain rather than lower extremity pain
* Subjects who are willing and capable of providing informed consent
* Subjects who are willing and capable of participating in all testing and questionnaire requirements associated with the clinical study

Exclusion Criteria:

* Any prior home use of the NexWave or any TENS/IFC device
* Any history of lumbar spine surgery or spinal fractures
* Subjects with a history of rheumatic disease
* Subjects with spine disorders, deformities, or severe spinal conditions such as scoliosis and kyphosis, Pott's disease, disc protrusion, or others that can be attributed to specific causes of back pain
* Subjects currently prescribed and adherent to opioid therapy
* Current implanted cardiac pacemakers, defibrillators, cardiac pumps, spinal stimulators, or other implanted electronic devices
* Active psychiatric or uncontrolled mood disorders including subjects on antipsychotic medication, diagnosis of bipolar disorder or schizophrenia, or uncontrolled anxiety or clinical depression
* Subjects with a known history of allergic reactions to medical adhesives or any condition that could affect placement of the electrodes
* Women of childbearing potential who are pregnant or who are planning to become pregnant during the anticipated study period
* Subjects with health conditions that in the Investigator's medical opinion would prevent participation in the study, interfere with assessment or therapy, significantly raise the risk of study participation, or modify outcome data or its interpretation
* Subjects who are currently enrolled in another investigational study that would directly interfere with the current study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale Pain Rating - NexWave vs. Sham | Four weeks
  VAS pain rating between baseline and four weeks for NexWave subjects as compared to sham device subjects.
Visual Analogue Scale Pain Rating - NexWave vs. Control | Four weeks
  VAS pain rating between baseline and four weeks for NexWave subjects as compared to control or sham device subjects.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) - NexWave vs. Sham | Four weeks
  ODI scores between baseline and four weeks for NexWave subjects as compared to sham device subjects.
Oswestry Disability Index (OD) - NexWave vs. Control | Four weeks
  ODI scores between baseline and four weeks for NexWave subjects as compared to control or sham device subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gilmore, MD, Principal Investigator — The Center for Clinical Research
Locations (8):
- United States (8):
  - DBPS Research, Greenwood Village, Colorado
  - McGreevy NeuroHealth, Saint Augustine, Florida
  - Peachtree Orthopedics, Atlanta, Georgia
  - Horizon Clinical Research, Jasper, Georgia
  - Applied Pain Institute, LLC, Bloomington, Illinois
  - One Oak Medical, Congers, New York
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - Summit Brain, Spine and Orthopedics, Lehi, Utah

IPD SHARING:
Plan to Share IPD: No